CLINICAL TRIAL: NCT05747846
Title: Intraoperative Pain in Carpal Tunnel Release Wide-awake Local Anesthesia With no Tourniquet vs Local Anesthesia With Tourniquet
Brief Title: Pain in Carpal Tunnel Release Wide-awake Local Anesthesia With no Tourniquet vs Local Anesthesia With Tourniquet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, IGNACIO RELLAN, Principal Investigator, Hospital Italiano de Buenos Aires
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5857
Record Dates: First submitted 2023-01-25; First posted 2023-02-28 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- wide-awake local anesthesia no tourniquet (Active Comparator): Patients will be operated under local anesthesia without a tourniquet (WALANT technique)
  Interventions: Procedure: Carpal tunnel release, WALANT technique
- Tourniquet (Active Comparator): Patients will be operated under local anesthesia with the use of a tourniquet
  Interventions: Procedure: Carpal tunnel release using a tourniquet

INTERVENTIONS:
Procedure: Carpal tunnel release, WALANT technique — Patients will receive 20 ml of 1% lidocaine with 1:100,000 epinephrine (buffered 10:1 with 8.4% sodium bicarbonate). Thirty minutes before carpal tunnel release surgery, 10 mL will be injected subcutaneously, and 10 mL will be injected into the carpal tunnel. Patients will go under open carpal tunnel release without a tourniquet.
  Arms: wide-awake local anesthesia no tourniquet
Procedure: Carpal tunnel release using a tourniquet — Patients will receive 20 ml of 1% lidocaine with 1:100,000 epinephrine (buffered 10:1 with 8.4% sodium bicarbonate). Thirty minutes before carpal tunnel release surgery, 10 mL will be injected subcutaneously, and 10 mL will be injected into the carpal tunnel. Patients will go under open carpal tunnel release using a hemostatic cuff. The hemostatic cuff will be insufflated at the level of the arm at a pressure of 100 mmHg higher than the patient's systolic pressure. The cuff will be removed once wound closure is complete.
  Arms: Tourniquet

SUMMARY:
The aim of this study is to compare pain, satisfaction, and experience between patients who underwent Carpal Tunnel Release with wide-awake local anesthesia no tourniquet technique and local anesthesia with a tourniquet.

DETAILED DESCRIPTION:
The surgical pathology of the hand has grown exponentially. In most cases, the resolution is performed in outpatients with short surgical times. Given the increased demand for this type of surgery, surgeons have sought different variables to reduce the costs and human resources. Thus, the wide-awake local anesthesia no tourniquet procedure (WALANT). It deals with the non-need for anesthetic monitoring and with the regional use of anesthesia with epinephrine.

Its use avoids placing a pneumatic cuff on the arm owing to the vasoconstrictive action of epinephrine. However, the drug takes 25-30 minutes to achieve the maximum hemostatic effect, and adverse effects, such as distal necrosis, have been reported.

Therefore, the technique of local anesthesia without epinephrine with a tourniquet (LA-T) is also used daily by hand surgeons.

The use of a tourniquet, a pneumatic cuff, for less than 20 minutes has been associated with the same or lower pain profiles than the wide-awake local anesthesia no tourniquet without running the risk of adverse effects of epinephrine.

The objective of this study is to compare and assess pain and patient experience after short-duration hand surgery using the WALANT and LA-T techniques. The investigators hypothesized that both types of procedures had a similar level of satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Carpal tunnel syndrome with surgical resolution
* Surgical procedures takes less than 30 minutes

Exclusion Criteria:

* Lost follow-up

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2023-08-07 (Actual); Study Completion 2023-08-26 (Actual)

PRIMARY OUTCOMES:
Pain during surgery | Immediately after surgery
  Visual analog scale. A numerical scale from 0 to 10 (a higher score means the worst outcome), where 0 indicates no pain, and 10 indicates the worst pain possible.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas M Molho, MD, Principal Investigator — Hospital Italiano de Buenos Aires
Locations (1):
- Hospital Italiano, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No